CLINICAL TRIAL: NCT02179437
Title: Retrospective Study to Investigate Intraoperative TIVA With Propofol on Postoperative Pain and Side Effects After Liver Resection Surgery
Brief Title: Intraoperative TIVA With Propofol on Postoperative Pain and Side Effects After Liver Resection Surgery
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Chi-Wai Cheung, Clinical Associate Professor, The University of Hong Kong
Other Study IDs: UW14-356
Record Dates: First submitted 2014-06-27; First posted 2014-07-01 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Postoperative Pain
Keywords: TIVA; Propofol; Postoperative pain; Liver resection surgery; Retrospective study
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Postoperative pain can be severe after liver resection surgery. However, postoperative pain management may be difficult for this group of patients. Opioidergic neurotransmission may be altered in cirrhotic patients and selectively increasing receptor affinity for opioids. Large dose of strong opioid may be required to achieve adequate pain control. However, this may not be possible due to the side effect of opioid and liver dysfunction after liver resection.

Propofol is a commonly used anaesthetic with rapid recovery and less side effects and TIVA (total intravenous analgesia) with propofol is a common technique now. The reduction on certain serum pro- inflammatory cytokines may lead to more smooth post- surgical recovery.

Recent case report proved the analgesic effect of propofol infusion. However other animal and clinical studies showed controversial result.

The aim of this retrospective study is to investigate the postoperative analgesic effects and side effects of intraoperative TIVA with propofol in patient undergoing liver resection surgery at Queen Mary Hospital, Hong Kong between 2010 to 2012.

DETAILED DESCRIPTION:
Retrospective audit.

Anaesthetic records and acute pain service records of patient undergone liver resection surgery between 2010 to 2012 in Queen Mary Hospital would be retrieved from the computer.

Data Collection

1. Demographic data;
2. Types of analgesic techniques;
3. Type of pain relief modalities;
4. Pain score up to 72 hours postoperatively;
5. Postoperative opioid consumption;
6. Incidence of adverse events during APS care;
7. Patients' satisfaction on pain relief.

Data Analysis For summarising analysis, mean or median with standard deviation or interquartile range will be reported. Parametric and non-parametric comparative tests will be used for analysis between/among patients with various characteristics. Kaplan Meier survival analysis and log-rank test will be used for duration of APS use.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergone liver resection surgery between 2010 to 2012 in Queen Mary Hospital

Exclusion Criteria:

* Essential data were missing.
* Patient participating in other research projects.
* Changes in postoperative pain management technique.
* Patients could not be assessed post-operatively for pain (i.e. post-operative IPPV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient undergone liver resection surgery between 2010 to 2012 in Queen Mary Hospital
Sampling Method: Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2016-02-22 (Actual); Study Completion 2016-02-22 (Actual)

PRIMARY OUTCOMES:
Postoperative pain score | From postoperative 1 hour to postoperative 72 hour

SECONDARY OUTCOMES:
Adverse event | From postoperative 1 hour to postoperative 72 hour

OTHER OUTCOMES:
Analgesic consumption | From postoperative 1 hour to postoperative 72 hour

CONTACTS AND LOCATIONS:
Overall Officials: Chi Wai Cheung, MD, Principal Investigator — Department of Anaesthesiology, The University of Hong Kong
Locations (1):
- Department of Anaesthesiology, The University of Hong Kong, Hong Kong, Hong Kong, China

REFERENCES:
- [Derived] Chan AC, Qiu Q, Choi SW, Wong SS, Chan AC, Irwin MG, Cheung CW. Effects of Intra-Operative Total Intravenous Anaesthesia with Propofol versus Inhalational Anaesthesia with Sevoflurane on Post-Operative Pain in Liver Surgery: A Retrospective Case-Control Study. PLoS One. 2016 Feb 22;11(2):e0149753. doi: 10.1371/journal.pone.0149753. eCollection 2016. PMID 26901037